CLINICAL TRIAL: NCT05948319
Title: The Effect of Myocardial Performance Index and Fetal Epicardial Thickness on Perinatal Outcomes in Obese Pregnant Women
Brief Title: the Fetal Epicardial Thickness in Obese Pregnant Women (EFT)
Acronym: EFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, şükran doğru, medical director, Necmettin Erbakan University
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Screening
Other Study IDs: 14221/neu
Record Dates: First submitted 2023-05-27; First posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Fetus Fetus; Pregnancy Complications
Keywords: obesity,; fetal epicardial thickness; myocardial performance index; perinatal outcome
MeSH Terms: conditions — Fetus-in-Fetu; Pregnancy Complications; Obesity | interventions — Ultrasonography, Doppler

STUDY DESIGN:
Intervention Model Description: case control
Who Masked: Participant
Masking Description: obese and non obese pregnant women
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- myocardial performance and epicard thickness in obese pregnant women (Active Comparator): obese pregnant versus normal-weight pregnant women were evaluated for MPI and fetal epicardial thickness
  Interventions: Diagnostic Test: Doppler ultrasonography
- obese pregnant (Active Comparator): obese pregnant versus normal-weight pregnant women were evaluated for MPI and fetal epicardial thickness
  Interventions: Diagnostic Test: Doppler ultrasonography

INTERVENTIONS:
Diagnostic Test: Doppler ultrasonography — Doppler study was performed in all cases. perinatal outcomes were evaluated.

SUMMARY:
the effects of fetal EFT on fetal cardiac function and fetal and maternal outcomes were investigated in obese pregnant women compared with normal-weight pregnant women.

DETAILED DESCRIPTION:
All pregnant women underwent a comprehensive fetal anomaly screening. One obstetrician (S.D.) assessed all of the measurements. Every measurement was performed using a convex 2-5 MHz Voluson E8 probe (GE Healthcare, Milwaukee, WI). Fetal biometry, UA, MCA Doppler, cerebroplacental ratio (CPR), modified MPI (mod-MPI), and EFT were assessed in accordance with the International Society of Ultrasound in Obstetrics and Gynecology (ISUOG) guidelines

ELIGIBILITY:
Inclusion Criteria:

* Obese pregnant women
* normal-weight pregnant women
* 24-40 gestational week

Exclusion Criteria:

Twin pregnancies, structural and chromosomal abnormalities, fetal rhesus isoimmunization, fetal growth restriction, cases with infections detected by maternal serological tests, pregestational or gestational diabetes (All patients underwent a 75-gram glucose load test at 24 weeks to rule out diabetes), preeclampsia, premature rupture of membranes were excluded from the study -

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
birth weight (gram) | birth 1 week
  fetal outcome
stillbirth rate (%) | birth 1 week
  fetal outcome
NICU admission | 6 months
  fetal outcome

CONTACTS AND LOCATIONS:
Overall Officials: şükran DR doğru, md, Study Director — NECMETTİN ERBAKAN UNIVERCITY; fatih dr akkuş, md, Principal Investigator — NECMETTİN ERBAKAN UNIVERCITY
Locations (1):
- Necmettin Erbakan University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
provided by the responsible researgher if requested
Supporting Information: CSR
Time Frame: 2 MONTHS
Access Criteria: VİA MAİL ADDRESS

REFERENCES:
- [Derived] Dogru S, Akkus F, Metin US, Acar A. Fetal Epicardial Fat Thickness in Obese Pregnant Women: Its Effect on Fetal Cardiac Function and Neonatal Outcomes. Z Geburtshilfe Neonatol. 2024 Oct;228(5):439-445. doi: 10.1055/a-2267-5478. Epub 2024 Mar 19. PMID 38503305